CLINICAL TRIAL: NCT04951674
Title: An Observational and Interventional Study on the Association Between Dietary Fibre and Cognitive Function in Healthy Volunteers
Brief Title: Dietary Fiber, Microbiota and Cognitive Function in Healthy Adults
Acronym: FOCUS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University College Cork (Other)
Responsible Party: Principal Investigator, John Cryan, Professor, University College Cork
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: APC135
Record Dates: First submitted 2021-06-08; First posted 2021-07-07 (Actual); Last update posted 2021-07-07 (Actual); Status verified 2021-07

CONDITIONS: Healthy
Keywords: Dietary fiber; Microbiota; Cognition; Diet; Microbiota-Gut-Brain Axis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DIET (Experimental): Participants will receive four individual, approximately 30-minute long dietary education sessions. The participants will receive detailed instructions (including meal plans, information on high fiber foods and serving sizes) on how to consume at least 30 grams of fiber per day.
  Interventions: Other: High fiber diet
- CONTROL (Placebo Comparator): No diet education. Group will spend same amount of time with study dietitian, but discussion is limited to review of current eating habits and minimal input on eating habits with referencing the standard food pyramid.
  Interventions: Other: Control diet

INTERVENTIONS:
Other: High fiber diet — 30 grams of fiber per day
  Arms: DIET
Other: Control diet — No diet education and change in diet
  Arms: CONTROL

SUMMARY:
Dietary fiber is well-known for its many health benefits, including the support of gastrointestinal, metabolic, and mental health. Although studies investigating whole dietary patterns in relation to cognition have demonstrated that diet quality and a healthy dietary pattern are associated with better cognitive performance, the role of dietary fiber in this regard is understudied. In the last decade, the role of the microbiota (trillions of microbes inhabiting the gut) in influencing various aspects of human health, including mental health and behavior, has also become established. Importantly, dietary fiber has been shown to positively affect the microbiota composition.

In this study, the role of dietary fiber in cognition through the lens of the microbiota is investigated. A two-part study including an observational (study 1) and interventional (study 2) arm has been designed. In study 1, the observational arm, 150 healthy individuals (30-60 years of age) will be recruited and grouped into high-fiber (>25 g/day, n=75) and low-fiber (<18 grams/day, n=75) consumers based on habitual dietary intake. Cognitive tasks (attention, episodic memory, decision making), psychological dimensions including impulsivity and emotional reactivity, biological samples (feces, blood, saliva, urine) and questionnaires about general health will be collected. In study 2, the interventional arm, a subgroup (n=60) of individuals from the low-fiber group will further be randomized into an 8-week randomized-controlled, parallel, single-blinded intervention to either receive a high fiber (n=30, aim 30 grams/day) or control (n=30) diet education. During the intervention period, individuals will provide repeated fecal samples in order to assess temporal microbial changes. At the end of the intervention period, individuals will undergo the same testing regarding cognitive and psychological variables and the same biological samples will be collected.

The investigators hypothesize that participants with higher dietary fiber intake at baseline will perform better in the cognitive tasks compared to individuals with low fiber intake, and that this difference can, in part, be mediated by the gut microbiota. Further the investigators hypothesize that through the dietary intervention the microbiota composition will positively shift to include more beneficial microbes and that cognitive performance will improve following the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Be able to give written informed consent.
* Be between 30 and 60 years of age.
* Be in generally good health as determined by the investigator.

Exclusion Criteria:

* Are less than 30 and greater than 60 years of age.
* Have a significant acute or chronic coexisting illness [cardiovascular, gastrointestinal (GI) [to include functional GI disorders, inflammatory bowel disease, celiac disease, lactose intolerance, food allergies], immunological, psychiatric [to include formal or as determined by MINI Psychiatric interview, diagnosis of current major depression, anxiety disorder, bipolar spectrum disorder, schizophrenia, other DSM-IV Axis I disorder], neurodevelopmental disorders, immunological, metabolic disorders [to include type I or II diabetes], or any condition which contraindicates, in the investigators judgement, entry to the study,
* Have a condition or taking a medication that the investigator believes would interfere with the objectives of the study, pose a safety risk or confound the interpretation of the study results; all psychoactive medications [to include anxiolytics, antipsychotics, antidepressants, anticonvulsants, centrally acting corticosteroids and opioid pain relievers), laxatives, enemas, antibiotics, anti-coagulants, over-the counter non-steroidal anti-inflammatories (NSAIDS). Participants should have a wash-out period of 4 weeks.
* Current prebiotic or probiotic supplement use (a wash-out period of 4 weeks after cessation will allow entry to the study).
* Females who are peri-menopausal, menopausal or post-menopausal.
* Females who are pregnant or planning a pregnancy, or lactating.
* Participants who are not fluent in English or English is not first language.
* Are color blind.
* Have dyslexia or dyscalculia.
* Are a current habitual daily smoker.
* Individuals who, in the opinion of the investigator, are considered to be poor attendees or unlikely for any reason to be able to comply with the trial.
* Participants receiving treatment involving experimental drugs. If the subject has been in a recent experimental trial, these must have been completed not less than 30 days prior to this study.
* Have a malignant disease or any concomitant end-stage organ disease.
* Have completed a study in the laboratory in the past 4 years.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-07 (Estimated); Primary Completion 2023-07 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Cognitive performance - Attention | Differences between groups at baseline and changes after 8-week of diet intervention in active group
  Assessment of attention using the Paced Auditory Serial Addition Test (PASAT)
Cognitive performance - Episodic memory | Differences between groups at baseline and changes after 8-week of diet intervention in active group
  Assessment of episodic memory using the Modified Rey Auditory Verbal Learning Test (ModRey)
Cognitive performance - Risky decision making | Differences between groups at baseline and changes after 8-week of diet intervention in active group
  Assessment of risky decision making using the Cambridge Gambling Task (CGT)
Cognitive performance - Affective decision making | Differences between groups at baseline and changes after 8-week of diet intervention in active group
  Assessment of affective decision making using the Iowa Gambling Task (IGT).

SECONDARY OUTCOMES:
Microbiota composition and function | Differences between groups at baseline and changes after 8-week of diet intervention in active group
  Shotgun sequencing of fecal samples
Blood inflammatory profile | Differences between groups at baseline and changes after 8-week of diet intervention in active group
  Cytokine and chemokine levels (e.g., TNFalpha, IL-10, IL-6) will be measured in lipopolysaccharide stimulated and unstimulated bloods
Salivary cortisol concentrations | Differences between groups at baseline and changes after 8-week of diet intervention in active group
  Morning cortisol awakening response
Stress assessment | Differences between groups at baseline and changes after 8-week of diet intervention in active group
  Perceived Stress Scale (range 0 to 40 with higher scores indicating higher perceived stress)
Anxiety assessment | Differences between groups at baseline and changes after 8-week of diet intervention in active group
  State Trait Anxiety Inventory (range 20-80 with higher scores indicating higher anxiety)
Emotion sensitivity, intensity, and persistence | Differences between groups at baseline and changes after 8-week of diet intervention in active group
  Emotion Reactivity Scale (range 0-84 with higher scores indicating higher dysfunctional emotional reactivity)
Impulsivity-related traits | Differences between groups at baseline and changes after 8-week of diet intervention in active group
  UPPS-P Impulsive Behavior Scale (range 59-236 with higher scores indicating higher dysfunctional impulsivity

CONTACTS AND LOCATIONS:
Overall Officials: John F Cryan, PhD, Principal Investigator — APC Microbiome Ireland, University College Cork; Gerard Clarke, PhD, Principal Investigator — APC Microbiome Ireland, University College Cork
Locations (1):
- APC Microbiome Ireland, University College Cork, Cork, Ireland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Berding K, Carbia C, Cryan JF. Going with the grain: Fiber, cognition, and the microbiota-gut-brain-axis. Exp Biol Med (Maywood). 2021 Apr;246(7):796-811. doi: 10.1177/1535370221995785. Epub 2021 Feb 28. PMID 33641478
- [Background] Cryan JF, O'Riordan KJ, Cowan CSM, Sandhu KV, Bastiaanssen TFS, Boehme M, Codagnone MG, Cussotto S, Fulling C, Golubeva AV, Guzzetta KE, Jaggar M, Long-Smith CM, Lyte JM, Martin JA, Molinero-Perez A, Moloney G, Morelli E, Morillas E, O'Connor R, Cruz-Pereira JS, Peterson VL, Rea K, Ritz NL, Sherwin E, Spichak S, Teichman EM, van de Wouw M, Ventura-Silva AP, Wallace-Fitzsimons SE, Hyland N, Clarke G, Dinan TG. The Microbiota-Gut-Brain Axis. Physiol Rev. 2019 Oct 1;99(4):1877-2013. doi: 10.1152/physrev.00018.2018. PMID 31460832